CLINICAL TRIAL: NCT04797221
Title: Development and Testing of a Veteran-Centered Lethal Means Safety Suicide Prevention Intervention (CDA 19-076)
Brief Title: Emergency Room Firearm and Medication Safety Intervention
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: CDX 21-003
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-07

CONDITIONS: Suicide; Firearm Injury; Overdose
Keywords: suicide
MeSH Terms: conditions — Suicide; Drug Overdose

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Veteran study group: The investigators will recruit approximately 20 Veterans who were identified as having elevated suicide risk while being treated in a VA Emergency Department.

SUMMARY:
Seventeen United States Veterans die by suicide each day. Nearly three-fourths of those Veterans die from firearm injury or poisoning, and many seek care in VA Emergency Departments (ED) prior to suicide attempts. In 2019, the VA began screening all Veterans seeking ED care for increased suicide risk. Interventions that promote firearm and medication safety are recommended for Veterans identified as at-risk. The investigators work will provide important information that will aid the development and testing of such an intervention for Veterans who seek care in VA EDs. The investigators will interview at-risk Veterans who recently sought VA ED care to identify factors relevant to developing the intervention, and work with Veterans and VA healthcare staff to develop and test an intervention.

DETAILED DESCRIPTION:
Veterans will be recruited from the Rocky Mountain Regional VA Medical Center (RMRVAMC) ED who are identified as having elevated suicide risk by VHA's new suicide risk screening initiative. All Veterans visiting VHA EDs are screened using an eight-item version of the Columbia Suicide Severity Rating Scale (C-SSRS) Screener, a valid predictor of future suicidal behavior. The C-SSRS Screener assesses suicide risk using eight items about recent suicidal ideation and intent, preparatory behaviors, and action. Deductive and inductive content analysis of qualitative interviews will occur in parallel with recruitment, and participants will be recruited until thematic saturation is achieved.

Veterans' visits (approx. 90 minutes) will be scheduled at their preferred times at RMRVAMC within two weeks of discharge from the ED. Sociodemographic and military service data will be collected using the Rocky Mountain Mental Illness Research, Education, and Clinical Center (MIRECC) Demographics Survey. During this visit, individuals will participate in qualitative interviews to identify contextual factors that may inform development of VA-based lethal means safety interventions.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* Recent Emergency Room care
* Screen positive for elevated suicide risk

Exclusion Criteria:

* Severe cognitive impairment
* Lack decisional capacity
* Unable to provide informed consent
* Lack reliable phone access
* Admitted to the hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans will be eligible who are seen for healthcare in the VA Emergency Department
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Simonetti, MD MPH, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (1):
- Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Group: 28 Veterans who were recently discharged from a VHA emergency care. Veteran participants were: >18 years of age, had access to firearms and/or medications at home, and were determined to be at elevated suicide risk based on the presence of suicide risk factors, including screening positive for having elevated suicide risk at the time of admission via the Columbia Suicide Severity Rating Scale Screener. Veterans were excluded if they were critically ill (intensive care unit requirements), are severely cognitively impaired, or had severe psychiatric symptoms that would preclude study participation.
Period: Overall Study
Arm/Group | Study Group
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Group
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (14.9)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Cisgender male | 24
  Gender: Cisgender female | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race / Ethnicity: African American / Black | 1
  Race / Ethnicity: White | 24
  Race / Ethnicity: Other | 2
  Race / Ethnicity: missing | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Qualitative Theme Among 28 Patients on Perspectives on Lethal Means Interventions
Description: Perspectives on VA-based interventions that aim to reduce access to firearms and medications.
Time Frame: baseline
Measure: Number; unit: participants
Arm/Group | Study Group
Number analyzed (Participants) | 28
participants
  Acceptability | 26
  Uncertainty about intent and efficacy | 20
  Cost and convenience are critical | 24
  Uncertainty regarding engaging other people in interventions | 14
  Influence of prior opioid exposure | 12

ADVERSE EVENTS:
Time Frame: 1 day
Description: this was not an intervention study and mortality was not assessed.
Arm/Group | Study Group
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-09): https://cdn.clinicaltrials.gov/large-docs/21/NCT04797221/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-05): https://cdn.clinicaltrials.gov/large-docs/21/NCT04797221/ICF_001.pdf